CLINICAL TRIAL: NCT04418921
Title: Self-Regulation in Children With Neurodevelopmental Disorders "SR-MRehab: Un Colegio Emocionante": a Protocol Study With Virtual Reality
Brief Title: Improving Self-regulation in Children With Neurodevelopmental Disorders:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Dulce Romero Ayuso, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR-MRehab
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Child Behavior Disorders; ASD; ADHD
MeSH Terms: conditions — Child Behavior Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Intervention on self-regulation will be carried out through a non-immersive virtual reality platform, "SR-Mrehab: Un colegio emocionante" in which students must conduct a series of activities designed specifically for this purpose. These activities will be performed by the children using mainly their hands to manage the virtual objects showed in the screen. To do this, our system make use of a Kinect motion sensor connected to the computer to control the body movements of the children. Moreover, our system records some relevant data of the execution of these activities for further analysis of the children's performance.The exercises will be divided into two blocks, emotional regulation (ER) and cognitive regulation (CR), in a total of 10 sessions, once a week, performing an exercise of each block per session. Each session will consists of 60 minutes. .
  Interventions: Behavioral: Self-regulation: MRehab - Un colegio emocionante, clinical trial with non-immersive virtual reality
- Control group (Active Comparator): The children from control group will follow a program of emotional education of Primary Schools, though group activities in the classroom (5, 49). Each session will last 50 minutes, just like in the experimental group. The content of the sessions will include 5 sessions of emotional awareness and 5 sessions of emotional and cognitive regulation. The activities are similar for the experimental group, but the virtual reality system will not be used. It will be held in parallel in another room of the school, on the same day and time, carried out by occupational therapists and students from the students in the last year of occupational therapy degree.
  Interventions: Behavioral: Traditional self-regulation program

INTERVENTIONS:
Behavioral: Self-regulation: MRehab - Un colegio emocionante, clinical trial with non-immersive virtual reality — The principles of the programme will be based on the following premises for children with ASD: 1) Strengthening communicative attempts; 2) Choose the most natural contexts possible; 3) Establish structured and predictable routines and environments; 4)Visually support information; 5) Adapting our language to the understanding level of the child. On the difficulty of interpreting and responding to social emotions and cues, games of perspectives are of great interest, where the child and therapist describe the same object from different perspectives, beliefs (guess that may be in this box), games with social stories, which are short stories that use pictograms, to help understand especially situations with social ambiguity: 1) describing what happens; 2) orienting the action, indicating to the child what to do in that situation; 3) anticipating and explaining what can happen and how you can feel; 4) developing a strategy that can be applied in similar situations.
  Arms: Experimental Group
Behavioral: Traditional self-regulation program — The children from control group will follow a program of emotional education of Primary Schools, though group activities in the classroom .The content of the sessions will include 5 sessions of emotional awareness and 5 sessions of emotional and cognitive regulation.Each session will last 50 minutes
  Other Names: Educative programa
  Arms: Control group

SUMMARY:
Children with neurodevelopmental disorders may show difficulties in self-regulation. The main objective of this study is to improve self-regulation skills in children between 6 and 11 years old with neurodevelopmental disorders. Methodology: A randomized controlled trial will be conducted with the use of "SF-MRehab: Un colegio emocionante", a non-inmersive virtual reality system where virtual objects can be managed by children in a natural way by using their hands. Children will be recruited from several schools from Granada (Spain) and they will be randomly allocated to two groups. Assessment will be conducted before and after the intervention as well as 24 weeks after the end of the intervention process. Experimental group will receive the intervention using virtual reality. Control group will receive the intervention through a standard self-regulation program. Both interventions will be performed once a week for a total of 10 sessions. Changes in self-regulation, as well as acceptability of technology with the use of SR-MRehab will be evaluated. The results will be published and will contribute with evidence regarding the use of this type of intervention on children with neurodevelopmental disorders

DETAILED DESCRIPTION:
The "SR-MRehab: un colegio Emocionante" is a randomized controlled trial, a non-inmersive virtual reality system will be conducted through Mrehab tool (39, 40). Children will be recruited from several schools from Granada (Spain) and they will be randomly allocated to two groups: experimental or control group. Assessment will be conducted before and after the intervention as well as 24 weeks after the end of the intervention process. Experimental group will receive the intervention using virtual reality. Control group will receive the intervention through a standard self-regulation program. Both interventions will be performed once a week for a total of 10 sessions (50 min sessions per day). The inclusion criteria are: 1) have special educational needs; 2) possible oral comprehension, with the possibility of fixing the gaze; 3) be able to attend to verbal and visual instructions; 4) maintain sustained attention for at least four minutes. Exclusion criteria are: 1) severe motor disability; 2) children with major behavioural problems, such as self-harm; 3) children with high abilities. Initially, all students of this center with special educational needs will be invited.

2.2. Procedure and Enrollment The implementation of the program covers the period from September 2019 to May 2020, divided into six stages: recruitment, pre-evaluation, assignation, intervention, post-evaluation and follow-up at 6 months. The initial stage corresponds to the acceptance by the management of the centers, and the subsequent invitation to the participants by sending a letter to the parents/legal guardians, which contains an informative document of the characteristics of the project and the corresponding informed consent for participate in it. Children are randomly assigned through the online randomization program. The type of allocation to each group will be by simple randomization. Recruitment and study procedure is shown in Figure 1 2.2.1. Study Variables The main variables of the study can be divided into two main dimensions: 1) executive functions: inhibitory control, flexibility, planning, reasoning, and problem solving; 2) socio-emotional competences: recognition of emotions, emotional regulation and social competence. These variables were and will be evaluated through several questionnaires provided to parents, teachers and students and test performed by children, as shown in Table 1.

Additionally, other sociodemographic data and information on the child's development and learning history were collected. Through the "SR-MRehab: un colegio emocionante", in each session, the following information will be collected for each task: number of hits, cognitive errors, time each participant to complete the task.

The assessment will be made in the first weeks of December 2020, dividing the assessment into three blocks. First, the EQ-i:YV questionnaire (41) and Clocks and Affect Recognition subtests from NEPSY-II (42) will be provided to students, and on the other hand, teachers and parents will asked to complete the EPYFEI-Escolar (44) and EPYFEI (45) questionnaires respectively, they'll have to fill in and come back within the next week. Second, the students will complete the assessment corresponding to the subtests of Design Fluency and Theory of Mind of the NEPSY-II. Finally, in a third session, they will carry out a final block to assess executive functions through Trail Making Test A and B (TMT A-B) and Stroop test.

The same evaluation will be carried out immediately after finishing the program. In addition, the acceptability of the technology will be evaluated with the children at the end of each session and at the end of the whole program. A combination of methods will be used to assess acceptability (46). Firsts, in each session, a visual analog scale will be used to evaluate each activity, type Smileyometer, which consists of a visual analog scale with coding based on a 5 point Likert scale (Horrible=1; Great=5). In addition, at the end of the program the method "This or That" will be used, though five questions, for example: what has been the most fun of the program? Or what game would you like to have at home?. To check the maintenance of the results of the program, a follow-up will be carried out at 3 months, in which the emotional regulation and executive functioning in the children will be re-assessed.

2.2.3. Intervention 2.2.3.1. Experimental Group Intervention on self-regulation will be carried out through a non-immersive virtual reality platform, "SR-Mrehab: Un colegio emocionante" in which students must conduct a series of activities designed specifically for this purpose. These activities will be performed by the children using mainly their hands to manage the virtual objects showed in the screen. To do this, our system make use of a Kinect motion sensor connected to the computer to control the body movements of the children. Moreover, our system records some relevant data of the execution of these activities for further analysis of the children's performance.

The exercises will be divided into two blocks, emotional regulation (ER) and cognitive regulation (CR), in a total of 10 sessions, once a week, performing an exercise of each block per session. Each session will consists of 60 minutes. In general, each session will take into account the development of the various executive functions: working memory, inhibitory control, flexibility, reasoning, planning and problem solving (15) and emotional competencies divided into the following dimensions: perception and emotional awareness, emotional regulation, emotional autonomy and social competence (47). Table 2 lists the organization, description and aims of each session. These sessions will take place from January to April 2021.

The MRehab tool allows establishing five levels of difficulty. Before starting the intervention program, a database will be created with each participant, assigning each of the tasks designed for each child according to the results of the previous assessment.

The intervention will begin with the explanation of the group session of 3 to 4 children. Subsequently, individually in order to record the responses and perform the activities, it will be asked to perform different tasks with the support and supervision of the occupational therapist and psychologist. The session would end with a small assembly in which each child discusses their experience and how and where the skills learned could be generalized in their activities of daily living. Each session will be one hour long.

2.2.3.2. Control Group

The children from control group will follow a program of emotional education of Primary Schools, though group activities in the classroom (5, 49). Each session will last 50 minutes, just like in the experimental group. The content of the sessions will include 5 sessions of emotional awareness and 5 sessions of emotional and cognitive regulation. The activities are similar as those listed in Table 2 for the experimental group, but the virtual reality system will not be used. It will be held in parallel in another room of the school, on the same day and time, carried out by occupational therapists and students from the students in the last year of occupational therapy degree.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Autism Spectrum Disorders and / or Attention Deficit Disorder with Hyperactivity
* Have special educational needs;
* Oral comprehension, with the possibility of fixing the gaze;
* Be able to attend to verbal and visual instructions;
* Be able to maintain sustained attention for at least four minutes.

Exclusion Criteria:

* Severe motor disability;
* Children with major behavioural problems, such as self-harm;
* Children with high abilities.

Initially, all students of this center with special educational needs will be invited.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Emotional Perception | 6 months
  Change in the number of errors in the recognition of recognized emotions on faces in the Affect Recognition subtest of the Children's Neuropsychology Assessment Battery (NEPSY-II), whose minimum scores are "0" and the maximum number of errors for children older than 6 years: 79. The higher the score, the worse the recognition of emotions.
Emotional Regulation | 6 months
  Change in the ability to understand mental functions, such as belief, intention, deceit, to understand the relationship between emotions and the social context, according to the Theory of Mind subtest of the Children's Neuropsychology Assessment Battery (NEPSY-II), whose minimum scores is "0" and the maximum score is 28. The higher the score, the better the ability to mentalize and recognize the mental states of other people.

SECONDARY OUTCOMES:
Cognitive Flexibility | 6 monhs
  Change in the skills of maintaining attention and for the ability to change and maintain a new pattern of responses, according to the Auditory attention and cognitive flexibility subtest of the Children's Neuropsychology Assessment Battery (NEPSY-II), whose minimum score is "0" and the maximum score is 30. The higher the score, the number of correct answers, the better the ability to attend and to be flexible with changes. In addition, it allows knowing the number of errors, divided into three types: commission, omission and inhibition errors. The greater the number of errors, the worse the attention and cognitive flexibility. The minimum error score is "0" and the maximum number of commission errors is 189, the maximum number of omission errors are 39, and the maximum number of inhibition errors is 33.
Planning, Sequencing | 6 months
  Change in planning and organization skills, as well as in self-supervision capacity, according to the Children's Neuropsychology Assessment Battery Clocks subtest (NEPSY-II), whose minimum scores are "0" and the maximum score is 78. A higher Score best ability to plan, sequence and monitor the action.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alcaniz ML, Olmos-Raya E, Abad L. [Use of virtual reality for neurodevelopmental disorders. A review of the state of the art and future agenda]. Medicina (B Aires). 2019;79(Suppl 1):77-81. Spanish. PMID 30776285
- [Background] Bashiri A, Ghazisaeedi M, Shahmoradi L. The opportunities of virtual reality in the rehabilitation of children with attention deficit hyperactivity disorder: a literature review. Korean J Pediatr. 2017 Nov;60(11):337-343. doi: 10.3345/kjp.2017.60.11.337. Epub 2017 Nov 27. PMID 29234356
- [Background] Parsons TD, Riva G, Parsons S, Mantovani F, Newbutt N, Lin L, Venturini E, Hall T. Virtual Reality in Pediatric Psychology. Pediatrics. 2017 Nov;140(Suppl 2):S86-S91. doi: 10.1542/peds.2016-1758I. PMID 29093039
- [Background] Eom H, Kim KK, Lee S, Hong YJ, Heo J, Kim JJ, Kim E. Development of Virtual Reality Continuous Performance Test Utilizing Social Cues for Children and Adolescents with Attention-Deficit/Hyperactivity Disorder. Cyberpsychol Behav Soc Netw. 2019 Mar;22(3):198-204. doi: 10.1089/cyber.2018.0377. Epub 2019 Jan 23. PMID 30672714
- [Result] Bekele E, Zheng Z, Swanson A, Crittendon J, Warren Z, Sarkar N. Understanding how adolescents with autism respond to facial expressions in virtual reality environments. IEEE Trans Vis Comput Graph. 2013 Apr;19(4):711-20. doi: 10.1109/TVCG.2013.42. PMID 23428456
- [Result] Voss C, Schwartz J, Daniels J, Kline A, Haber N, Washington P, Tariq Q, Robinson TN, Desai M, Phillips JM, Feinstein C, Winograd T, Wall DP. Effect of Wearable Digital Intervention for Improving Socialization in Children With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Pediatr. 2019 May 1;173(5):446-454. doi: 10.1001/jamapediatrics.2019.0285. PMID 30907929
- [Result] Bekele E, Crittendon J, Zheng Z, Swanson A, Weitlauf A, Warren Z, Sarkar N. Assessing the utility of a virtual environment for enhancing facial affect recognition in adolescents with autism. J Autism Dev Disord. 2014 Jul;44(7):1641-50. doi: 10.1007/s10803-014-2035-8. PMID 24419871
- [Result] Yuan SNV, Ip HHS. Using virtual reality to train emotional and social skills in children with autism spectrum disorder. London J Prim Care (Abingdon). 2018 Jun 7;10(4):110-112. doi: 10.1080/17571472.2018.1483000. eCollection 2018. PMID 30083244
- [Result] Shema-Shiratzky S, Brozgol M, Cornejo-Thumm P, Geva-Dayan K, Rotstein M, Leitner Y, Hausdorff JM, Mirelman A. Virtual reality training to enhance behavior and cognitive function among children with attention-deficit/hyperactivity disorder: brief report. Dev Neurorehabil. 2019 Aug;22(6):431-436. doi: 10.1080/17518423.2018.1476602. Epub 2018 May 17. PMID 29771624
- [Result] Blume F, Hudak J, Dresler T, Ehlis AC, Kuhnhausen J, Renner TJ, Gawrilow C. NIRS-based neurofeedback training in a virtual reality classroom for children with attention-deficit/hyperactivity disorder: study protocol for a randomized controlled trial. Trials. 2017 Jan 24;18(1):41. doi: 10.1186/s13063-016-1769-3. PMID 28118856
- [Derived] Romero-Ayuso D, Alcantara-Vazquez P, Almenara-Garcia A, Nunez-Camarero I, Trivino-Juarez JM, Ariza-Vega P, Molina JP, Gonzalez P. Self-Regulation in Children with Neurodevelopmental Disorders "SR-MRehab: Un Colegio Emocionante": A Protocol Study. Int J Environ Res Public Health. 2020 Jun 12;17(12):4198. doi: 10.3390/ijerph17124198. PMID 32545534